CLINICAL TRIAL: NCT06830460
Title: Efficacy of a Theoretical-practical Course for the Ultrasound Measurement of the Optic Nerve Diameter in Different Healthcare Operators
Brief Title: Measurement of the Optic Nerve Diameter in Different Healthcare Operators
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Associate Professor in Anesthesia and Intensive Care Medicine, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ONSD
Record Dates: First submitted 2025-02-06; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer; Healthy Volunteer Study
Keywords: optic nerve sheath diameter; theoretical-practical course

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ONSD training (Experimental)
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — The training will consist of a four-hour session, including a 30-minute lecture on ocular anatomy and ultrasound techniques, a real-time demonstration, and supervised hands-on practice with at least 20 measurements.
  Participants must achieve a score of at least 70% on a multiple-choice test to proceed to practical verification, where they will measure the ONSD in five healthy volunteers. These measurements will be compared to those taken by an expert tutor.

SUMMARY:
The study evaluates the effectiveness of a theoretical-practical training course for the ultrasound measurement of the optic nerve sheath diameter (ONSD), a non-invasive method used to estimate intracranial pressure (ICP). The optic nerve sheath is continuous with the subarachnoid space, which contains cerebrospinal fluid (CSF). An increase in ICP leads to an increase in CSF within the sheath, enlarging its diameter. ONSD measurement is typically performed by placing an ultrasound probe on the closed eyelid, allowing visualization of the optic nerve behind the eyeball.

While the correlation between ONSD enlargement and elevated ICP is well-documented, there is variability in diagnostic cut-off values due to differences in measurement techniques, equipment, and operator experience. Previous studies have shown that even novice operators can achieve clinically acceptable accuracy after brief training.

This study aims to assess whether medical students, nursing students, anesthesiology and intensive care residents, and intensive care nurses can learn to perform reliable ONSD measurements after a short training session.

Methodology:

The study will involve 40 participants unfamiliar with ONSD measurement: 10 medical students, 10 nursing students, 10 anesthesiology and intensive care residents, and 10 experienced intensive care nurses. The training will consist of a four-hour session, including a 30-minute lecture on ocular anatomy and ultrasound techniques, a real-time demonstration, and supervised hands-on practice with at least 20 measurements.

Participants must pass a multiple-choice test with at least 70% correct answers to proceed to practical verification, where they will measure ONSD in five healthy volunteers. These measurements will be compared with those taken by an expert tutor.

Measurement Technique:

The ultrasound technique follows expert consensus guidelines, using a linear probe with a minimum frequency of 7.5 MHz. Volunteers will be positioned semi-seated at a 45° head elevation with closed eyelids. The ONSD measurement will be taken 3 mm behind the retina on the right eye. Care will be taken to avoid pressure on the eyeball, and safety parameters will be monitored to ensure compliance with FDA guidelines.

The study aims to demonstrate that various healthcare professionals can achieve accurate and reliable ONSD measurements with proper training, enhancing the utility of this technique in diverse clinical settings.

DETAILED DESCRIPTION:
INTRODUCTION The measurement of the optic nerve sheath diameter (ONSD) is a non-invasive diagnostic technique used to estimate intracranial pressure (ICP). The optic nerve sheath, which surrounds the optic nerve, is continuous with the subarachnoid space, which contains cerebrospinal fluid (CSF). When ICP increases, the amount of cerebrospinal fluid in the optic nerve sheath also increases, causing an enlargement of its diameter.

The measurement of ONSD is performed non-invasively using ultrasound by placing an ultrasound probe on the closed eyelid to visualize the optic nerve behind the eyeball [3]. Guidelines on how to measure ONSD have recently been published in a statement by an international consensus of experts.

The correlation between increased ONSD and elevated ICP is well documented. An ONSD exceeding reference values can indicate elevated intracranial pressure. Although it is not a continuous monitoring method, ONSD measurement can be performed repeatedly at the patient's bedside and in remote locations without causing significant discomfort to the operator or patient, which may be invaluable for patient triage and management. It can also be useful for the continuous assessment of critically ill patients in tertiary care centers, especially those too unstable to be transported to the radiology department for a CT scan or MRI.

The diagnostic cut-off values indicating elevated ICP vary across studies and meta-analyses. Generally, reported values range between 4.8 mm and 6.4 mm. This variability is influenced by several factors, including measurement techniques, equipment used, and operator experience.

To date, no clear and direct data demonstrate that healthcare professionals other than medical specialists (with varying levels of expertise) can learn this technique and obtain reliable ONSD measurements. Therefore, we designed this study to assess the ability of medical students, nursing students, anesthesiology and intensive care residents, and intensive care nurses to visualize and correctly measure ONSD in healthy volunteers after a brief training course on the technique.

MATERIALS AND METHODS

The study will be conducted in the classrooms of the "Magna Graecia" University of Catanzaro after approval by the local ethics committee. Written informed consent will be obtained from all participants. The trial will be prospectively registered on clinicaltrials.gov.

Subjects

A total of 40 participants naive to the ONSD measurement technique will be recruited as follows:

* 10 medical students
* 10 nursing students
* 10 anesthesiology and intensive care medicine residents
* 10 intensive care nurses with at least 3 years of experience

Training Session All participants will attend a theoretical-practical training session of approximately four hours based on current literature, focusing on the key principles of the technique, including acoustic windows and anatomical landmarks for ONSD measurement.

The session will include a 30-minute lecture covering the anatomy of the eyeball and orbit, ultrasound technique, and ONSD measurement. A real-time demonstration of how to obtain ONSD measurements will follow. Participants will then perform at least 20 supervised ONSD measurements under the guidance of an expert tutor to familiarize themselves with the ultrasound procedure and reduce intra- and inter-observer variability. At the end of the session, each participant will have the opportunity to perform five additional examinations if they do not yet feel confident.

Verification Session All participants will take a multiple-choice questionnaire consisting of 10 questions. A score of at least 70% will be required to pass. Those who pass the theoretical test will proceed to the practical assessment.

In the practical assessment, each participant will perform ONSD measurements on five healthy volunteers who were not involved in the training session. These measurements will be recorded and compared to the reference measurement performed by the expert tutor.

ONSD Measurement Technique The technique presented to trainees and subsequently applied for measurement follows the recent expert consensus on quality criteria for ONSD evaluation. Operators will use an ultrasound machine equipped with an ocular ultrasound preset and a linear probe with a minimum effective frequency of 7.5 MHz.

Healthy volunteers will be positioned semi-seated with a 45° head elevation, maintaining a neutral gaze with closed eyelids. The image will be acquired by centering the eyeball within the frame in an axial plane and adjusting the ultrasound beam to insonate the optic nerve perpendicularly. Once the image is sufficiently clear to distinguish anatomical structures without artifacts, it will be captured for ONSD measurement. The measurement will be taken 3 mm posterior to the retina, considering the internal diameter of the ONSD. Since the volunteers are healthy and have no neurological pathology, only the right ONSD will be measured in all subjects.

The obtained measurement will be recorded by an external researcher. Throughout all scans, operators will be reminded to avoid applying pressure to the eyeball. Additionally, volunteers will be repeatedly asked to report any discomfort or pressure beyond a gentle touch on the eyes during each measurement. This ensures both safety and measurement accuracy, as excessive pressure on the eyeball could cause eye injury and/or increase intraocular pressure.

Although an ocular preset will be used, considering the potentially prolonged scan time, safety parameters set by the Food and Drug Administration (FDA) will be monitored and maintained, specifically a thermal index <1 and a mechanical index <0.23. The probe will be properly cleaned and disinfected between each measurement.

During the entire measurement procedure, the expert tutor will note any execution errors using a specially designed checklist.

ELIGIBILITY:
Inclusion Criteria:

* medical student, or nurse student, or residents in anesthesia or nurse with at least 3 years of Intensive care unit experience

Exclusion Criteria:

* previous skills on ONSD measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
OSND measure affidability | Through study completion, an average of 3 hours
  ONSD measure will be recorded and compared to that one from a expert tutor

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- Magna Graecia University, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
pseudonymised data will be share on reasonable request to the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after study pubblication
Access Criteria: On reasonable request for scientific purposes

REFERENCES:
- [Background] Potgieter DW, Kippin A, Ngu F, McKean C. Can accurate ultrasonographic measurement of the optic nerve sheath diameter (a non-invasive measure of intracranial pressure) be taught to novice operators in a single training session? Anaesth Intensive Care. 2011 Jan;39(1):95-100. doi: 10.1177/0310057X1103900116. PMID 21375098
- [Background] Soliman I, Johnson GGRJ, Gillman LM, Zeiler FA, Faqihi F, Aletreby WT, Balhamar A, Mahmood NN, Ahmad Mumtaz S, Alharthy A, Lazaridis C, Karakitsos D. New Optic Nerve Sonography Quality Criteria in the Diagnostic Evaluation of Traumatic Brain Injury. Crit Care Res Pract. 2018 Apr 30;2018:3589762. doi: 10.1155/2018/3589762. eCollection 2018. PMID 29854448
- [Background] Hirzallah MI, Lochner P, Hafeez MU, Lee AG, Krogias C, Dongarwar D, Hartman ND, Ertl M, Robba C, Malojcic B, Valaikiene J, Sarwal A, Hakimi R, Schlachetzki F; Optic Nerve Sheath Diameter Point-of-Care Ultrasonography Quality Criteria Checklist (ONSD POCUS QCC) Expert Panelists. Optic Nerve Sheath Diameter Point-of-Care Ultrasonography Quality Criteria Checklist: An International Consensus Statement on Optic Nerve Sheath Diameter Imaging and Measurement. Crit Care Med. 2024 Oct 1;52(10):1543-1556. doi: 10.1097/CCM.0000000000006345. Epub 2024 Jun 5. PMID 38836697
- [Background] Geeraerts T, Launey Y, Martin L, Pottecher J, Vigue B, Duranteau J, Benhamou D. Ultrasonography of the optic nerve sheath may be useful for detecting raised intracranial pressure after severe brain injury. Intensive Care Med. 2007 Oct;33(10):1704-11. doi: 10.1007/s00134-007-0797-6. Epub 2007 Aug 1. PMID 17668184
- [Background] Liu D, Kahn M. Measurement and relationship of subarachnoid pressure of the optic nerve to intracranial pressures in fresh cadavers. Am J Ophthalmol. 1993 Nov 15;116(5):548-56. doi: 10.1016/s0002-9394(14)73195-2. PMID 8238213